CLINICAL TRIAL: NCT03249766
Title: Prospective Observational Study of Prevalence of Ipsilateral Shoulder Pain in Patients After Thoracic Surgeries
Brief Title: Study of Prevalence of Ipsilateral Shoulder Pain in Patients After Thoracic Surgeries
Status: Completed | Type: Observational
Sponsor: Tata Memorial Hospital (Other Government)
Responsible Party: Principal Investigator, Raghu Thota, Associate Professor, Tata Memorial Hospital
Other Study IDs: 1900
Record Dates: First submitted 2017-08-10; First posted 2017-08-15 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational — Observational study

SUMMARY:
Thoracic surgeries are associated with significant operative trauma1. While thoracic epidural analgesia may help control the incisional component of the pain, an excruciating postthoracotomy. Ipsilateral Shoulder Pain (ISP) could under mine pain management in the post thoracotomy patient2. The incidence of ISP ranges from 21% to 97%3. ISP impairs respiration, mobility, and physical therapy in the early postoperative period4. The etiology of ISP is unclear. Several hypotheses have been proposed as possible causes of ISP, including transection of a major bronchus, ligament distraction by surgical retraction, shoulder joint strain as a result of intraoperative positioning, pleural irritation due to the thoracostomy tube, and referred pain from irritation of the pericardium or mediastinal and diaphragmatic surfaces2, 5, 6. ISP is defined as the pain occurring on the operated side of thoracic surgeries in the immediate postoperative period as early as one hour after surgery6,of dull aching, stabbing, burning, electric or throbbing nature of moderate to severe intensity and resistant to treatment, most commonly located in the region of the deltoid muscle or on the posterior or superior surface of the arm or above ⅓ of the lateral part of the clavicle on the anterior surface of the chest, lasting 3-4 days2, 7-11.The primary objective of this study is to find out the prevalence of ISP and the risk factors associated with it.

DETAILED DESCRIPTION:
This will be a prospective observational study, which will be done over a period of one year (Upto 250 patients) after approval from ethics committee. The data of the first three months will be analysed (Upto 60 patients) and will presented as a thesis for MD (Anaesthesia). It will be carried out at Tata Memorial Centre, Mumbai. After Institutional Ethics Committee approval, Written informed consent in the language the patient understands the best will be obtained undergoing thoracic surgeries where the pleura is opened including Thoracotomy, Video Assisted Thoracic Surgeries (VATS). Data over a three months period will be collected. Pain at the incisional site and Ipsilateral shoulder pain (ISP) will be assessed separately using the numeric rating scale (NRS) during the patients' stay in the postanesthesia care unit (PACU) by an independent assessor, at 1 hour, 6 hours and 12 hours after coming to the PACU. The characteristics, intensity and pain at shoulder at rest and movement will also be assessed. Data including age, sex, BMI, American Society of Anesthesiologists (ASA) physical status, diagnosis, side and type of operation, surgical approach, positioning during surgery, duration of surgery, type of regional anesthesia, and, in patients with epidural anesthesia, level of catheter placement will also be recorded.

All male & female patients (aged 18-75 years) who undergo thoracic surgeries where the pleura is opened including Video Assisted Thoracic Surgeries (VATS)

EXCLUSION CRITERIA:

1. presence of preoperative shoulder pain,
2. preoperative shoulder pathology,
3. use of analgesics for more than 1 week preoperatively,
4. inability to understand the numeric rating scale(NRS)scoring system for pain assessment
5. failure to extubate at the end of surgery.
6. Patients who haven't given consent
7. Age < 18yrs and > 75 yrs.

STATISTICAL ANALYSIS:

Since the study will be done over a period of twelve months, there is no sample size.

Continuous variables will be analyzed using independent t-test or Mann Whitney U test as per the distribution of the data for continuous variables. Categorical variables will be analyzed using Chi-square test or Fisher's exact test. P-value < 0.05 will be considered statistical significant. Risk factors of ISP will be analyzed using univariate and multivariate binary regression with robust estimates to calculate odds ratio (OR) and their 95% confidence interval. A manual stepwise forward logistic regression will be used to extract univariate independent variables. A p value ≤ 0.2 by univariate analysis will be used as the criterion for choosing variables to be included in the model for multivariate analysis. A p value <0.05 is considered statistically significant. Cut-off points of the independent variables, including age group and duration of surgery, are estimated by the method of maximum likelihood to achieve best discrimination between patients with and without ISP.

ELIGIBILITY:
Inclusion Criteria:

* All male & female patients (aged 18-75 years) who undergo thoracic surgeries where the pleura is opened including Video Assisted Thoracic Surgeries (VATS)

Exclusion Criteria:

* presence of preoperative shoulder pain,
* preoperative shoulder pathology,
* use of analgesics for more than 1 week preoperatively,
* inability to understand the numeric rating scale(NRS)scoring system for pain assessment
* failure to extubate at the end of surgery.
* Patients who haven't given consent
* Age < 18yrs and > 75 yrs.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This will be a prospective observational study, which will be done over a period of one year (Upto 250 patients) after approval from ethics committee. The data of the first three months will be analysed (Upto 60 patients) and will presented as a thesis for MD (Anaesthesia). It will be carried out at Tata Memorial Centre, Mumbai. Data over a three months period will be collected. Pain at the incisional site and Ipsilateral shoulder pain (ISP) will be assessed separately using the numeric rating scale (NRS) during the patients' stay in the postanesthesia care unit (PACU) by an independent assessor, at 1 hour, 6 hours and 12 hours after coming to the PACU. The characteristics, intensity and pain at shoulder at rest and movement will also be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 370 (Actual)
Dates: Start 2017-08-22 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
Prevalence of Ipsilateral shoulder pain | Upto 12 hours post surgery
  Numeric rating scale within 12 hours post operative

CONTACTS AND LOCATIONS:
Overall Officials: Raghu S Thota, MD, Principal Investigator — Tata Memorial Hospital
Locations (1):
- Tata Memorial Centre, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided